CLINICAL TRIAL: NCT05136092
Title: A Pilot Study to Determine Fructose Uptake by Primary Human Colorectal Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 21-03023487
Record Dates: First submitted 2021-11-11; First posted 2021-11-26 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Tumors
Keywords: Fructose; D-Xylose; Primary Human Colorectal Tumors
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fructose

STUDY DESIGN:
Intervention Model Description: Prospective, pilot, feasibility, single-center, non-randomized, open-label, phase 1, investigator-initiated study to evaluate the specific uptake of fructose by human colorectal tumors with 12 subjects in 2 cohorts:
  Cohort 1: fructose-fed with 6 subjects Cohort 2: xylose-fed with 6 subjects.
  Eligible subjects scheduled to undergo colorectal resection for cancer treatment will be invited to participate in the study in consecutive order from the practice of colorectal surgeons at the time of their preoperative clinic visit. First, Cohort 1 subjects will be enrolled followed by the Cohort 2 subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: HFCS (fructose-fed) (Experimental): On the day of Surgery, between two and three hours before surgery.
  Subjects will prepare the sugar solutions (Fructose-containing solution: 250 mL of water containing 41.25 g of D-Fructose and 33.75 g of D-Glucose) by adding 250 ml water to the sugar powder provided by the study team and drink it between two and three hours before surgery. Subjects will be reminded the day before the surgery to drink the solution.
  Interventions: Dietary Supplement: Cohort 1: HFCS (fructose) fed
- Cohort 2: D-Xylose (xylose-fed) (Experimental): On the day of Surgery, between two and three hours before surgery.
  Subjects will prepare the sugar solutions (Xylose-containing solution: 250 mL of water containing 41.25 g of D-Xylose and 33.75g of D-Glucose) by adding 250 ml water to the sugar powder provided by the study team and drink it betweentwo and three hours before surgery. Subjects will be reminded the day before the surgery to drink the solution.
  Interventions: Dietary Supplement: Cohort 2: D-Xylose (xylose-fed)

INTERVENTIONS:
Dietary Supplement: Cohort 1: HFCS (fructose) fed — Two to three hours before surgery. Subjects will prepare the sugar solutions (Fructose-containing solution: 250 mL of water containing 41.25 g of D-Fructose and 33.75 g of D-Glucose) by adding 250 ml water to the sugar powder provided by the study team and drink it between two and three hours before surgery.
  Samples collected before surgery:
  * Blood sample of 5 ml
  * Urine Samples 5 ml
  Day of Surgery The anesthesia and surgical procedure will undergo as per regular care. Samples collection at the time the surgical specimen is removed
  * Blood sample of 5 ml blood will be obtained from the IV line
  * Tissue samples
    * 2 Tumor tissue samples 5mmx5mmx5mm,
    * 2 Intestinal /colon tissue samples 5mmx5mmx5mm
    * 2 tissue samples from mesentery tissue 5mmx5mmx5mm
  * Optional Liver Biopsy - a 3-5 mm liver tissue will be obtained for research.
  * Urine Samples 5 ml
  Arms: Cohort 1: HFCS (fructose-fed)
Dietary Supplement: Cohort 2: D-Xylose (xylose-fed) — Two to three hours before surgery.
  Subjects will prepare the sugar solutions (Xylose-containing solution: 250 mL of water containing 41.25 g of D-Xylose and 33.75g of D-Glucose) by adding 250 ml water to the sugar powder provided by the study team and drink it between two and three hours before surgery.
  Samples collected before surgery:
  * Blood sample of 5 ml
  * Urine Samples 5 ml
  Day of Surgery The anesthesia and surgical procedure will undergo as per regular care. Samples collection at the time the surgical specimen is removed
  * Blood sample of 5 ml blood will be obtained from the IV line
  * Tissue samples
    * 2 Tumor tissue samples 5mmx5mmx5mm,
    * 2 Intestinal /colon tissue samples 5mmx5mmx5mm
    * 2 tissue samples from mesentery tissue 5mmx5mmx5mm
  * Optional Liver Biopsy - a 3-5 mm liver tissue will be obtained for research.
  * Urine Samples 5 ml
  Arms: Cohort 2: D-Xylose (xylose-fed)

SUMMARY:
This proposed study is designed to investigate the specific uptake of fructose by human colorectal tumors. In this study, subjects with colorectal cancer undergoing surgery will receive an oral sugar solution containing fructose or xylose prior to surgery. The tumor will then be resected, and a portion of the tissue will be used to measure the abundance of fructose and xylose. The study hypothesis is that the tumors will take up fructose sugar but not xylose sugar. A comparison of the sugar uptake between the tumor and normal tissues from the adjacent intestinal epithelium and smooth muscle and the liver will be conducted. This proposal will confirm that human colorectal cancer tumors can directly absorb dietary sugars, which has never been demonstrated.

DETAILED DESCRIPTION:
This prospective pilot study is designed to investigate the uptake of dietary fructose and xylose by primary human colon tumors. In this study, the recruited patients with colorectal cancer will receive an oral sugar solution containing either Fructose sugar or Xylose sugar before surgery. The tumor will then be resected and a portion of the tumor, normal intestinal tissue, blood, urine, and liver will be used to quantify fructose and xylose.

* Research question Can primary human tumors take up fructose or xylose?
* A statement of the hypothesis The hypothesis is that fructose, but not xylose, can be directly absorbed and stored by primary human colon tumors.
* Design Prospective, non-randomized, pilot, feasibility, single-center, open-label, phase 1, investigator-initiated study to evaluate the uptake of dietary fructose and xylose by primary human colon tumors with 12 subjects in 2 cohorts: Cohort 1: 6 subjects will consume a sugar solution containing fructose and Cohort 2: 6 subjects will consume a sugar solution containing xylose. Eligible subjects that are scheduled to undergo colorectal resection for cancer treatment will be invited to participate in the study in consecutive order from the practice of colorectal surgeons at the time of their preoperative clinic visit. First, Cohort 1 subjects will be enrolled followed by the Cohort 2 subjects.

N=12 Subjects Cohort 1: Fructose sugar solution =6 Subjects Cohort 2: Xylose sugar solution=6 Subjects

ELIGIBILITY:
Inclusion Criteria:

* Subjects of 18 years of age or older, male, and female
* Subjects with a diagnosis of invasive non-hereditary colonic adenocarcinoma who will be undergoing standard of care (SOC) laparoscopic, robot-assisted, or open surgical resection
* The subject provides informed consent

Exclusion Criteria:

* Subjects with a history of uncontrolled diabetes mellitus (A1C >7.0) Type I and Type 2, will be excluded to avoid potential confounders associated with the consumption of a large bolus of sugar (e.g., hyperglycemia and hyperinsulinemia)
* Inflammatory Bowel Disease (Ulcerative Colitis or Crohn's Disease)
* Patients on steroid medications
* Patients with current infectious disease
* Subjects who do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
The abundance of fructose in tumor extracts | Morning after the consumption of oral sugar solutions(during surgery at the time of specimen removal)
  The abundance of fructose in tumor extracts assessed by mass spectrometry in the morning after the consumption of oral sugar solutions.

SECONDARY OUTCOMES:
The abundance of Fructose and [13C]-Fructose in the blood | Morning after the consumption of oral sugar solutions(during surgery at the time of specimen removal)
  The abundance of Fructose and [13C]-Fructose in the blood in the morning after the consumption of oral sugar solutions assessed by mass spectrometry.
Abundance of Fructose and [13C]-Fructose in the urine | Morning after the consumption of oral sugar solutions(during surgery at the time of specimen removal)
  The abundance of Fructose and [13C]-Fructose in the urine in the morning after the consumption of oral sugar solutions assessed by mass spectrometry.
Abundance of Fructose and [13C]-Fructose in the liver | Morning after the consumption of oral sugar solutions(during surgery at the time of specimen removal)
  The abundance of Fructose and [13C]-Fructose in the liver tissue in the morning after the consumption of oral sugar solutions assessed by mass spectrometry.
Abundance of Fructose and [13C]-Fructose in the intestine | Morning after the consumption of oral sugar solutions(during surgery at the time of specimen removal)
  The abundance of Fructose and [13C]-Fructose in the intestine tissue in the morning after the consumption of oral sugar solutions assessed by mass spectrometry.
Abundance of Fructose and [13C]-Fructose in the mesentery tissues | Morning after the consumption of oral sugar solutions(during surgery at the time of specimen removal)
  The abundance of Fructose and [13C]-Fructose in the mesentery tissue in the morning after the consumption of oral sugar solutions assessed by mass spectrometry.
The abundance of Xylose and [13C]-Xylose in the blood | Morning after the consumption of oral sugar solutions(during surgery at the time of specimen removal)
  The abundance of Xylose and [13C]-Xylose in the blood in the morning after the consumption of oral sugar solutions assessed by mass spectrometry.
The abundance of Xylose and [13C]-Xylose in the urine | Morning after the consumption of oral sugar solutions(during surgery at the time of specimen removal)
  The abundance of Xylose and [13C]-Xylose in the urine in the morning after the consumption of oral sugar solutions assessed by mass spectrometry.
The abundance of Xylose and [13C]-Xylose in the liver | Morning after the consumption of oral sugar solutions(during surgery at the time of specimen removal)
  The abundance of Xylose and [13C]-Xylose in the liver tissue in the morning after the consumption of oral sugar solutions assessed by mass spectrometry.
The abundance of Xylose and [13C]-Xylose in the intestinal tissue | Morning after the consumption of oral sugar solutions(during surgery at the time of specimen removal)
  The abundance of Xylose and [13C]-Xylose in the intestinal tissue in the morning after the consumption of oral sugar solutions assessed by mass spectrometry.
The abundance of Xylose and [13C]-Xylose in the mesentery tissues | Morning after the consumption of oral sugar solutions(during surgery at the time of specimen removal)
  The abundance of Xylose and [13C]-Xylose in the mesentery tissues in the morning after the consumption of oral sugar solutions assessed by mass spectrometry.
The abundance of Xylose and [13C]-Xylose in the in the tumor | Morning after the consumption of oral sugar solutions(during surgery at the time of specimen removal)
  The abundance of Xylose and [13C]-Xylose in the tumor in the morning after the consumption of oral sugar solutions assessed by mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Mehraneh D Jafari, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No